CLINICAL TRIAL: NCT07353684
Title: Phase II Clinical Study of Adebrelimab Plus Apatinib and SOX Regimen for Conversion Therapy of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Adebrelimab, Apatinib & SOX for Conversion Therapy in Advanced Gastric/GEJ Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, DengWei, Chief Physician, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFHHS20250003; BFHHS20250003 (Registry Identifier: Beijing Friendship Hospital, Capital Medical University)
Record Dates: First submitted 2025-03-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Adebrelimab; Adenocarcinoma of GE Junction; Adenocarcinoma of Stomach
Keywords: adebrelimab; Adenocarcinoma of GE junction; Adenocarcinoma of stomach; conversion therapy
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab + Apatinib + SOX (Experimental): Participants receive Adebrelimab, Apatinib, Oxaliplatin, and S-1 as conversion therapy. Treatment is administered in 3-week cycles for 2-8 cycles, followed by surgical assessment.
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: Adebrelimab — 1200 mg, iv.gtt, single infusion, 21 days as a cycle, Day 1
Drug: Apatinib — 250mg, p.o, qd, 21 days as a cycle
Drug: SOX Chemotherapy — Oxaliplatin: 130mg/m2, iv.gtt, single infusion, 21 days as a cycle, Day 1. Tigio: 40mg (body surface area(BSA)<1.25m2), 50mg (BSA≥1.25m2, and BAS<1.5m2), 60mg (BSA ≥1.5m2), p.o, bid, 21 days as a cycle, Day 1-14.

SUMMARY:
This is a prospective, single-center, single-arm, open phase II clinical study. Forty-nine participants with pathologically or cytologically confirmed gastric cancer or gastroesophageal junction cancer are scheduled to be enrolled in this study. All participants will be treated with 2 to 8 cycles of adebrelimab, apatinib, oxaliplatin, and tigio before surgery. Participants will evaluate the treatment effect after every 2 cycles of medication. By the investigator assessment as an operable subject, apatinib was discontinued for one cycle. The adjuvant treatment will be determined by the investigators based on the participants' postoperative pathology results. Participants requiring adjuvant therapy, with a postoperative interval of at least 4 weeks, but not more than 10 weeks. When the resection standard isn't met for 8 cycles of treatment, the treatment is switched to a maintenance phase, which the subject treatment regimen is determined by the investigator. During the treatment period, participants will receive the study drugs on Day 1 of each 21-day cycle until evidence of disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Study Design: This is a prospective, single-center, single-arm, open-label Phase II clinical study. The study aims to evaluate the efficacy and safety of Adebrelimab combined with Apatinib and SOX regimen as conversion therapy for patients with advanced, unresectable gastric or gastroesophageal junction (GEJ) adenocarcinoma. The study plans to enroll approximately 49 participants who are assessed by investigators as having conversion therapy potential (defined as single organ metastasis, retroperitoneal lymph node metastasis, supraclavicular lymph node metastasis, limited peritoneal metastasis, or invasion of surrounding organs).

Treatment Protocol: Eligible participants will receive a four-drug combination therapy consisting of Adebrelimab, Apatinib Mesylate, Oxaliplatin, and S-1. The treatment is administered in 3-week cycles:

Adebrelimab: 1200 mg, intravenous infusion on Day 1.

Apatinib Mesylate: 250 mg, oral, once daily.

Oxaliplatin: 130 mg/m², intravenous infusion on Day 1.

S-1 (Tegafur, Gimeracil, and Oteracil Potassium): 40-60 mg (based on Body Surface Area), oral, twice daily on Days 1-14.

Study Procedures and Phases:

Conversion Treatment Phase: Patients will receive treatment for a minimum of 2 cycles and a maximum of 8 cycles. Resectability will be assessed by the investigator every 2 cycles using imaging evaluation.

Surgical Intervention:

If the tumor is assessed as resectable: Apatinib will be discontinued for one cycle prior to the planned surgery to ensure safety.

Surgery should be performed between 3 to 6 weeks (maximum 6 weeks) after the last dose of the study drug.

Post-operative Phase: The decision to administer adjuvant therapy will be made by the investigator based on post-operative pathological results. If adjuvant therapy is required, it will commence at least 4 weeks but no later than 10 weeks after surgery.

Maintenance Phase: If the tumor remains unresectable after 8 cycles of combination therapy, the patient will transition to a maintenance phase. The specific treatment regimen during the maintenance phase will be determined by the investigator based on the patient's condition.

Follow-up: Upon discontinuation of treatment, patients will undergo safety follow-ups every 30 days until 90 days after the last dose. Subsequently, patients will enter the survival follow-up period to monitor disease recurrence, metastasis, and overall survival. Follow-ups will occur every 3 months for the first 2 years and every 6 months for years 2 to 5.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years at the time of enrollment, with an estimated life expectancy of ≥ 3 months.
* Histologically or cytologically confirmed gastric cancer or gastroesophageal junction cancer, predominantly adenocarcinoma.
* Unresectable locally advanced gastric or gastroesophageal junction adenocarcinoma (Stage III or IV), as determined by the investigator based on CT, MRI, and/or PET-CT.
* Disease with conversion (translational) therapeutic potential, as assessed by the investigator.
* No prior anti-tumor treatment, including chemotherapy, radiotherapy, targeted therapy, immunotherapy, or other systemic anticancer therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate hematologic function within 14 days prior to enrollment:

  * White blood cell count ≥ 3.5 × 10⁹/L.
  * Absolute neutrophil count ≥ 1.5 × 10⁹/L.
  * Hemoglobin ≥ 90 g/L (9.0 g/dL).
  * Platelet count ≥ 100 × 10⁹/L.
  * Adequate hepatic function within 14 days prior to enrollment:Total bilirubin ≤ 1.5 × upper limit of normal (ULN);ALT and AST ≤ 2.5 × ULN in patients without liver metastases;ALT and AST ≤ 5 × ULN in patients with liver metastases;Adequate renal function:Serum creatinine ≤ 1.5 × ULN;Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment and agree to use effective contraception during the study and for at least 12 weeks after the last dose.
* Male participants must be surgically sterile or agree to use effective contraception during the study and for at least 12 weeks after the last dose
* Ability to understand and willingness to sign a written informed consent form
* Expected to comply with study procedures and follow-up requirements

Exclusion Criteria:

* HER2-positive gastric or gastroesophageal junction adenocarcinoma.
* Conditions that may significantly affect oral drug absorption, including inability to swallow, persistent nausea or vomiting, chronic diarrhea, or intestinal obstruction.
* Known hypersensitivity or allergy to adebrelimab, apatinib, oxaliplatin, S-1 (tegafur/gimeracil/oteracil), or any of their excipients.
* History of severe allergic reactions to monoclonal antibodies.
* Active autoimmune disease or autoimmune disorders requiring systemic treatment.
* Congenital or acquired immunodeficiency.
* Use of systemic immunosuppressive therapy within 14 days prior to the first dose of study treatment.
* Administration of live attenuated vaccines within 4 weeks prior to the first dose or planned during the study period.
* Severe infection within 4 weeks prior to initiation of study treatment.
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Evidence of interstitial lung disease, including pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonitis, or severely impaired pulmonary function.
* Uncontrolled hypertension despite at least 3 months of antihypertensive treatment.
* Uncontrolled clinically significant cardiovascular disease.
* High risk of severe bleeding, as judged by the investigator.
* Peripheral neuropathy of Grade > 2 according to CTCAE.
* Participation in another interventional clinical trial within 4 weeks prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
* Any condition that, in the investigator's judgment, makes the participant unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-05-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | At the time of definitive surgery following completion of neoadjuvant treatment (within 6 months from enrollment)
  Proportion of participants who achieve R0 resection, defined as microscopically margin-negative resection confirmed by postoperative pathological examination.
Adverse Events (AE) | From treatment initiation to 30 days after the last dose of study treatment (up to approximately 6 months).
  Incidence, nature, and severity of treatment-emergent adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 1year
  ORR is defined as the percentage of participants who achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | Up to 3 years
  Time from day of study to death due to any cause.
Disease Free Survival (PFS) | Up to 2 years
  Time from enrollment to disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No